CLINICAL TRIAL: NCT04575142
Title: Comparison of Office-based KTP and CO2 Laser Outcomes in Patients With Vocal Cord Lesions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01463
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Laryngeal Diseases
MeSH Terms: conditions — Laryngeal Diseases | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO2 laser device group (Experimental): Participants who will be undergoing laser treatment for their vocal nodes with a specific laser device. AcuPulse Duo, a CO2 laser is absorbed by water found in soft tissues and is independent of tissue color. It is very precise and causes less damage of the deep tissues, which results in less swelling and faster recovery. The absence of a long healing process means that most patients can resume their normal activities even on the same day The CO2 laser is the preferred laser for use in the operating room.
  Interventions: Device: CO2 laser

INTERVENTIONS:
Device: CO2 laser — the CO2 laser (AcuPulse DUO, Lumenis, Yokneam, Israel) generally ranges from 3 to 10 W in superpulse mode, with 0.05 second on/0.01 second off, depending on lesion size and location of the lesion(s).
  The CO2 laser can be used in a continuous, pulsed, or superpulsed mode. The superpulsed mode reduces the exposure time to a few nanoseconds while delivering high energies of 400 to 500 W with each peak. The rest time between each peak allows the tissues to cool and reduces thermal injury to adjacent tissues.
  Other Names: AcuPulse Duo

SUMMARY:
The purpose of this study is to test the outcomes of a CO2 laser device called AcuPulse Duo on vocal lesions and compare them to the most commonly used Aura KTP laser in order to determine which device has the best results. The CO2 laser device is an already FDA approved device. However, there have been no studies comparing the two devices for this use.

DETAILED DESCRIPTION:
A flexible laryngoscope is passed through the patient's nose. Energy from the laser is delivered through a fiber. This unique quality allows the physician to thread the fiber through an endoscope and deliver energy. KTP is uniquely effective because the laser uses green light, which has an affinity with blood vessels. This means that the energy from the laser is absorbed more easily by blood vessels than other tissue. Targeting the blood supply of a lesion causes the lesion to slough off, leaving the surrounding tissue undamaged. However, the properties of the KTP are not necessarily ideal, in that it penetrates deep into the vocal fold, risking scar formation. On the other hand, the CO2 laser is absorbed by water found in soft tissues and is independent of tissue color. It is very precise and causes less damage of the deep tissues, which results in less swelling and faster recovery. The absence of a long healing process means that most patients can resume their normal activities even on the same day The CO2 laser is the preferred laser for use in the operating room. The purpose of the study is to evaluate the fiber-based version of the CO2 laser in the office setting.

ELIGIBILITY:
Inclusion Criteria:

* Presence of laryngeal papillomatosis, hemorrhagic polyps, or leukoplakia/dysplasia of the vocal folds requiring in-office treatment.
* Has the capacity to provide consent

Exclusion Criteria:

* Accutane (Isotretinoin) within the past 6-12 months
* History of keloid formation
* Demonstration of excessive or unusually prolonged erythema

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in mucosal wave grade | Treatment Visit (Day 0), Follow up Visit (6-12 weeks)
  Absolute change from baseline in mucosal wave grade using videostroboscopy on each treated vocal fold 2-3 months after the treatment for both groups. Videostroboscopy is a standard of care procedure for patients with voice problems and would be performed regardless of the subject's participation in the study.
Absolute and percentage change from baseline | Treatment Visit (Day 0), Follow up Visit (6-12 weeks)
  Absolute and percentage change from baseline in the Voice Handicap Index (VHI) score 2-3 months after the treatment. Measured by Voice Handicap Index (VHI-10), a self reported questionnaire assessing the frequency of characteristics of their voice and the effects their voice has on their lives. 10 statements using a scale where 0 is "Never" and 4 is "Always"
Change in Physician's satisfaction | Treatment Visit (Day 0), Follow up Visit (6-12 weeks)
  In using a self reported questionnaire to determine how easy it was to use the CO2 laser. Questions asked: Ease of use, completeness of treatment, bleeding issues, complications and case time from laser start to finish.
Change in Patient's discomfort | Treatment Visit (Day 0), Follow up Visit (6-12 weeks)
  Patient comfort during the procedure will be measured by Patient Discomfort questionnaire. (All lesion types). The Patient-Comfort Scale is a 5 scale rating: 1- no, 2- minimal, 3-mild, 4-moderate, 5-severe.
Change in Lesion regression | Treatment Visit (Day 0), Follow up Visit (6-12 weeks)
  Lesion regression (based on endoscopic measurement technique) Stills from the laryngoscopic exam will be imported and measured into the Image J software.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Amin, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to achlae01@nyu.edu. To gain access, data requestors will need to sign a data access agreement.